CLINICAL TRIAL: NCT01321957
Title: FOLFOX and Bevacizumab With or Without Irinotecan in First-line Treatment for Metastatic Colorectal Cancer. A Randomized Phase II Study
Brief Title: Efficacy of FOLFOX+Bevacizumab in Combination With Irinotecan in the Treatment of Metastatic Colorectal Cancer
Acronym: CHARTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Hans-Joachim Schmoll, MD, MD, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-0209
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Bevacizumab; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOX+Bevacizumab (Active Comparator): bevacizumab at a dose of 5 mg/kg iv over 30 to 90 min (day 1) oxaliplatin at a dose of 85 mg/m2 iv over two hours (day 1) I-LV at a dose of 200 mg/m2 iv over two hours (day 1) 5-FU at a dose of 3200 mg/ m2 iv over 48 hours (day 1-3)
  Interventions: Drug: Oxaliplatin, 5FU/LV, Bevacizumab
- FOLFOX+Bevacizumab+Irinotecan (Experimental): bevacizumab at a dose of 5 mg/kg iv over 30 to 90 min (day 1) irinotecan at a dose of 165 mg/m2 iv over two hours (day 1) oxaliplatin at a dose of 85 mg/m2 iv over two hours (day 1) I-LV at a dose of 200 mg/m2 iv over two hours (day 1) 5-FU at a dose of 3200 mg/ m2 iv over 48 hours (day 1-3)
  Interventions: Drug: 5FU/LV, Oxaliplatin, Bevacizumab, Irinotecan

INTERVENTIONS:
Drug: Oxaliplatin, 5FU/LV, Bevacizumab — bevacizumab at a dose of 5 mg/kg iv over 30 to 90 min (day 1) oxaliplatin at a dose of 85 mg/m2 iv over two hours (day 1) I-LV at a dose of 200 mg/m2 iv over two hours (day 1) 5-FU at a dose of 3200 mg/ m2 iv over 48 hours (day 1-3)
  Other Names: Bevacizumab; Oxaliplatin; I-LV; 5-FU
  Arms: FOLFOX+Bevacizumab
Drug: 5FU/LV, Oxaliplatin, Bevacizumab, Irinotecan — bevacizumab at a dose of 5 mg/kg iv over 30 to 90 min (day 1) irinotecan at a dose of 165 mg/m2 iv over two hours (day 1) oxaliplatin at a dose of 85 mg/m2 iv over two hours (day 1) I-LV at a dose of 200 mg/m2 iv over two hours (day 1) 5-FU at a dose of 3200 mg/ m2 iv over 48 hours (day 1-3)
  Other Names: Bevacizumab; Oxaliplatin; I-LV; 5-FU; Irinotecan
  Arms: FOLFOX+Bevacizumab+Irinotecan

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Irinotecan in combination with FOLFOX+Bevacizumab versus FOLFOX+Bevacizumab alone in the first-line treatment of patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
5-Fluorouracil and oxaliplatin (FOLFOX-Regimen) in combination with bevacizumab is regarded as standard first-line treatment in metastatic colorectal cancer [Saltz et al., 2008]. Current studies established the role of the FOLFOXIRI regimen [Souglakos et al., 2006, Falcone et al., 2007]. A further intensification of the therapy seems feasible yielding response rates up to 84% and a disease control rate up to 100% [Falcone, 2008, Santomaggio, 2009, Masi, 2010]. This trial evaluates the activity of an intensified first-line therapy for metastatic colorectal cancer compared to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed diagnosis of stage IV (UICC) colorectal cancer (primary tumor may be present)
2. Patients with at least one measurable lesion, with size > 1 cm (RECIST v1.1)
3. ECOG Performance status ≤ 2 (ECOG 2, only if tumor related)
4. Patients, who are able to tolerate intensive first lien treatment as judged by the investigator
5. Life expectancy > 3 months
6. Age ≥ 18 years
7. Haematologic function: ANC ≥ 1.5 x 109/L, platelets ≥ 100 x109/L, hemoglobin

   * 9 g/dl or 5.59 mmol/l
8. Patients not receiving therapeutic anticoagulation must have an INR < 1.5 ULN and aPTT < 1.5 ULN within 7 days prior to registration. The use of full dose anticoagulants is allowed as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least two weeks at the time of registration.
9. Adequate liver function as measured by serum transaminases (AST & ALT) ≤ 2.5 x ULN (in case of liver metastases < 5 x ULN) and total bilirubin ≤ 1.5 x ULN
10. Adequate renal function: Serum creatinine ≤ 1.5 x ULN
11. Signed, written informed consent

Exclusion Criteria:

1. Patients with histologically confirmed diagnosis of stage IV (UICC) colorectal cancer (primary tumor may be present)
2. Patients with at least one measurable lesion, with size > 1 cm (RECIST v1.1)
3. ECOG Performance status ≤ 2 (ECOG 2, only if tumor related)
4. Patients, who are able to tolerate intensive first lien treatment as judged by the investigator
5. Life expectancy > 3 months
6. Age ≥ 18 years
7. Haematologic function: ANC ≥ 1.5 x 109/L, platelets ≥ 100 x109/L, hemoglobin

   * 9 g/dl or 5.59 mmol/l
8. Patients not receiving therapeutic anticoagulation must have an INR < 1.5 ULN and aPTT < 1.5 ULN within 7 days prior to registration. The use of full dose anticoagulants is allowed as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least two weeks at the time of registration.
9. Adequate liver function as measured by serum transaminases (AST & ALT) ≤ 2.5 x ULN (in case of liver metastases < 5 x ULN) and total bilirubin ≤ 1.5 x ULN
10. Adequate renal function: Serum creatinine ≤ 1.5 x ULN
11. Signed, written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
progression free survival rate | 9 months after first study drug administration

SECONDARY OUTCOMES:
tumour response according to RECIST v 1.1 | until progression of disease for a maximum of two years after end of treatment
Secondary resection rate | for a maximum of two years after end of treatment
Progression free survival rate | until progression of disease for a maximum of two years after end of treatment
Overall survival | until death for a maximum of two years after end of treatment
Adverse events | 18 months after the date of last study drug administration
  Toxicity of study medication
Quality of Life evaluated by questionnaire | Until end of treatment (maximum 2 years after first study drug administration)
  Quality of Life evaluated using questionnaire EORTC QLQ-30

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joachim Schmoll, MD, Principal Investigator — Universitätsklinikum Halle
Locations (51):
- Germany (51):
  - Medizinische Klinik mit Schwerpunkt Hämatologie und Onkologie, Berlin
  - Knappschaftskrankenhaus Bottrop, Bottrop
  - Onkologische Praxis, Bottrop
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Cologne
  - Studiengesellschaft Kátay + Reiser GbR, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - Evangelisches Krankenhhaus Dinslaken, Dinslaken
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Onkozenrum Dresden, Dresden
  - Onkologie Duisburg, Duisburg
  - St. Georg Klinikum Eisenach gGmbH, Eisenach
  - Katholisches Krankenhaus St. Johann Nepomuk, Erfurt
  - pioh Praxis, Frechen
  - Partnerschaft FÄ für Innere Medizin, Freiberg
  - MVZ Osthessen GmbH, Fulda
  - Kreiskrankenhaus Gummersbach GmbH, Gummersbach
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Marienkrankenhaus Hamburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Überörtliche Gemeinschaftspraxis für Innere Medizin, Hamburg
  - Klinikum Region Hannover GmbH,, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Praxis Dr. Schröder, Hanover
  - Klinikum Heidenheim, Heidenheim
  - SP Hämatologie u. Internistische Onkologie, Hennigsdorf
  - Onkologische Schwerpunktpraxis im Medicinum, Hildesheim
  - St. Bernward Krankenhaus, Hildesheim
  - Sanaklinikum Hof GmbH, Hof
  - Institut für med. Dokumentation, Gutachtenerstellung, Gesundheitsförderung u. Qualitätssicherung GbR, Kaiserslautern
  - St. Cincentius-Kliniken gAG, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Praxis für Innere Medizin und Gastroenterologie, Köthen
  - Praxis für Innere Medizin, Laatzen
  - Ortenau Klinikum - Lahr Ettenhaim, Lahr
  - Gemeinschaftspraxis Dr. med. Veling-Kaiser, Landshut
  - Medizinisches Versorgungszentrum Mitte, Leipzig
  - Onco Studies Lörrach-OSL an der Schwerpunktpraxis Onkologie Dreiländereck, Loerrach
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Universitätsklinikum Magdeburg, Magdeburg
  - Internistisches Fachzentrum mit Dialyse, Onkologische Praxis am Klinikum, Memmingen
  - Friedrich-Ebert-Krankenhaus Neumünster GmbH, Neumünster
  - PIUS-Hospital Oldenburg, Oldenburg
  - Universitätsklinikum Rostock, Rostock
  - MedResearch - Medizinisches Studien- u. Dokumentationszentrum Leipziger Land, Rötha
  - Praxis für Innere Medizin, Hämatololgie und Onkologie, Schkeuditz
  - Leopoldina Krankenhaus der Stadt Schweinfurt GmbH, Schweinfurt
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - Praxisnetzwerk Hämaologie/Intern. Onkologie, Troisdorf
  - Ammerland-Klinik GmbH, Westerstede
  - Praxisgemeinschaft für Onkologie und Urologie Wilhelmshaven, Wilhelmshaven
  - Praxis Dr. med. Mathias Schulze, Zittau

REFERENCES:
- [Derived] Schmoll HJ, Mann J, Meinert F, Garlipp B, Borchert K, Vogel A, Goekkurt E, Kaiser U, Hoeffkes HG, Russel J, Kanzler S, Edelmann T, Forstbauer H, Gohler T, Hannig C, Hildebrandt B, Roll C, Bokemeyer C, Steighardt J, Cygon F, Ibach S, Stein A, Tintelnot J. Efficacy and quality of life for FOLFOX/bevacizumab +/- irinotecan in first-line metastatic colorectal cancer-final results of the AIO CHARTA trial. Br J Cancer. 2024 Feb;130(2):233-241. doi: 10.1038/s41416-023-02496-4. Epub 2023 Nov 23. PMID 37996507
- [Derived] Cremolini C, Antoniotti C, Stein A, Bendell J, Gruenberger T, Rossini D, Masi G, Ongaro E, Hurwitz H, Falcone A, Schmoll HJ, Di Maio M. Individual Patient Data Meta-Analysis of FOLFOXIRI Plus Bevacizumab Versus Doublets Plus Bevacizumab as Initial Therapy of Unresectable Metastatic Colorectal Cancer. J Clin Oncol. 2020 Aug 20:JCO2001225. doi: 10.1200/JCO.20.01225. Online ahead of print. PMID 32816630
- [Derived] Stein A, Glockzin G, Wienke A, Arnold D, Edelmann T, Hildebrandt B, Hollerbach S, Illerhaus G, Konigsrainer A, Richter M, Schlitt HJ, Schmoll HJ. Treatment with bevacizumab and FOLFOXIRI in patients with advanced colorectal cancer: presentation of two novel trials (CHARTA and PERIMAX) and review of the literature. BMC Cancer. 2012 Aug 16;12:356. doi: 10.1186/1471-2407-12-356. PMID 22897915